CLINICAL TRIAL: NCT03877601
Title: A Prospective Follow-up Intervention Study: Detection of Early Esophageal Cancer by Near-infrared Fluoresence Molecular Endoscopy Using Bevacizumab-800CW
Brief Title: Detection of Early Esophageal Cancer by NIR-FME.
Acronym: ESCEND
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Collaborators: Helmholtz Zentrum München (Industry)
Responsible Party: Principal Investigator, dr. W.B. Nagengast, MD, Principal investigator, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL68582.042.18
Record Dates: First submitted 2019-02-27; First posted 2019-03-15 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Barrett Esophagus
Keywords: Fluorescence; Endoscopy; Bevacizumab-800CW
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Topical administration of bevacizumab-800CW (Experimental): The tracer will be topically administered 5 minutes prior to the fluorescence endoscopy procedure (with the near infrared fluorescence endoscopy platform).
  Interventions: Drug: Bevacizumab-IRDye800CW; Diagnostic Test: Fluorescence endoscopy

INTERVENTIONS:
Drug: Bevacizumab-IRDye800CW — Topical administration of Bevacizumab-IRDye800CW during the endoscopic procedure.
Diagnostic Test: Fluorescence endoscopy — Device: Molecular Fluorescence Endoscopy platform A flexible fluorescence fiber-bundle is attached to a fluorescence camera platform to enable the detection of fluorescence signals. The fluorescence fiber-probe is inserted through the standard working channel of the standard clinical endoscope.

SUMMARY:
To improve detection of esophageal (pre)malignant lesions during surveillance endoscopy of patients at risk of developing malignancies, for example in Barrett's Esophagus (BE), there is a need for better endoscopic visualization and the ability for targeted biopsies. Optical molecular imaging of neoplasia associated biomarkers could form a promising technique to accommodate this need. It is known that the biomarker Vascular Endothelial Growth Factor (VEGF) is overexpressed in dysplastic and neoplastic areas in BE segments versus normal tissue and has proven to be a valid target for molecular imaging. The University Medical Center Groningen (UMCG) developed a fluorescent tracer by labeling the VEGF-targeting humanized monoclonal antibody bevacizumab, currently used in anti-cancer therapy, with the fluorescent dye IRDye800CW. The phase I study, named VICE, completed within the UMCG, showed that synchronal use of VEGFA-guided near-infrared fluorescence molecular endoscopy (NIR-FME) and high-definition white light endoscopy (HD-WLE), following topical or systemic tracer administration, could be practiced to recognize dysplastic and early EAC lesions in patients with BE. Furthermore, early lesion detection was improved by ~33% using the topically applied tracer approach compared with HD-WL/NBI endoscopy. With this phase 2 intervention study the investigators aim to statistically confirm previous pilot (Phase I) clinical data showing that the combination of HD-WLE and FME using labelled bevacizumab improves early EC detection over the current clinical standard.

DETAILED DESCRIPTION:
See brief summary

ELIGIBILITY:
Inclusion Criteria:

* Suspicion or diagnosed LGD, HGD or superficial EAC and planned diagnostic and/or therapeutic endoscopy.
* Age: 18 years or older.
* Written informed consent.

Exclusion Criteria:

* Patients younger than 18 years old
* Submucosal and invasive EAC; EAC with TNM-classification other than T1.
* Radiation therapy for esophageal cancer
* Immunoglobulin allergy
* Chemotherapy, immunotherapy or surgery 28 days before administration of the tracer
* Prior Bevacizumab treatment
* Non-adjustable hypertension
* Medical or psychiatric conditions that compromise the patient's ability to give informed consent.
* Pregnancy or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-07-29 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Fluorescence signal in patients with Barrett's Esophagus | During the endoscopic procedure
  Evaluating the performance of FME with topical administration of Bevacizumab-800CW for detection of neoplasia in BE patients compared to HD-WLE to make an estimation of the diagnostic accuracy in terms of sensitivity and specificity in order to make a power size calculation for the Phase III trial.

SECONDARY OUTCOMES:
Ex vivo fluorescence singals | 2 years
  Correlate and validate fluorescence signals detected in vivo with ex vivo histopathology grade of dysplasia and VEGF expression
Number of participants with adverse events (AE), serious adverse events (SAE) and suspected unexpected serious adverse reactions (SUSAR). | Up to 1 week after administration of tracer
  Data collection as a measure of safety and tolerability regarding administration of Bevacizumab-IRDye800CW
Interrogate potential new EC biomarkers | 2 years
  We will perform ex-vivo binding experiments with tracers against GREM1, -SULF1 and -PRKCi on the fresh EMR if available and compare them against the in-vivo WLE/NIR-FME findings. We will analyze the sensitivity and specificity of the novel markers alone or in combination. The targeting moieties will be coupled with different fluorophores allowing for multi-parametric analysis.

CONTACTS AND LOCATIONS:
Overall Officials: W.B. Nagengast, MD, PhD, PharmD, Principal Investigator — University Medical Center Groningen; Vasilis Ntziachristos, Prof. Dr., Principal Investigator — Helmholtz Zentrum München
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nagengast WB, Hartmans E, Garcia-Allende PB, Peters FTM, Linssen MD, Koch M, Koller M, Tjalma JJJ, Karrenbeld A, Jorritsma-Smit A, Kleibeuker JH, van Dam GM, Ntziachristos V. Near-infrared fluorescence molecular endoscopy detects dysplastic oesophageal lesions using topical and systemic tracer of vascular endothelial growth factor A. Gut. 2019 Jan;68(1):7-10. doi: 10.1136/gutjnl-2017-314953. Epub 2017 Dec 15. No abstract available. PMID 29247063